CLINICAL TRIAL: NCT00076024
Title: Randomized, Placebo-Controlled, Double-Blind, Phase 2 Study Of AG-013736 In Combination With Docetaxel Versus Docetaxel Alone In Patients With Metastatic Breast Cancer Preceded By A Phase 1 Evaluation Of The Combination
Brief Title: AG-013736 In Combination With Docetaxel Versus Docetaxel Alone For Patients With Metastatic Breast Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A4061010
Record Dates: First submitted 2004-01-12; First posted 2004-01-14 (Estimated); Results first posted 2012-03-16 (Estimated); Last update posted 2012-06-26 (Estimated); Status verified 2012-06

CONDITIONS: Breast Neoplasms
Keywords: metastatic breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Docetaxel; Axitinib

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Docetaxel + Placebo (Other): Docetaxel + Placebo
  Interventions: Drug: Placebo; Drug: Docetaxel
- Docetaxel + AG-013736 (Experimental): Docetaxel + AG-013736
  Interventions: Drug: AG-013736 (axitinib); Drug: Docetaxel

INTERVENTIONS:
Drug: Placebo — 5 mg twice daily [bid] continuous dosing
  Arms: Docetaxel + Placebo
Drug: Docetaxel — Standard of care drug administration
  Arms: Docetaxel + Placebo
Drug: AG-013736 (axitinib) — 5mg twice daily [bid] continuous dosing
  Arms: Docetaxel + AG-013736
Drug: Docetaxel — Standard of care drug administration
  Arms: Docetaxel + AG-013736

SUMMARY:
The primary purpose of the study is to determine the time to progression of the combination of study drug (AG-013736) and docetaxel versus docetaxel alone in patients who have not received prior chemotherapy for metastatic breast cancer. The secondary purpose of the study is to determine the dose of study drug that can be given with docetaxel administered on an every 3 week schedule.

ELIGIBILITY:
Inclusion Criteria:

* Female patients with histologically/cytologically proven metastatic breast carcinoma (stage IV, or recurrent with local or regional spread or distant metastatic disease)
* Adequate bone marrow, liver, and renal function

Exclusion Criteria:

* Adjuvant chemotherapy given in the past 12 months
* Uncontrolled brain metastases

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 174 (Actual)
Dates: Start 2004-02; Primary Completion 2007-01 (Actual); Study Completion 2008-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (46):
- United States (20):
  - Pfizer Investigational Site, Tucson, Arizona
  - Pfizer Investigational Site, Berkeley, California
  - Pfizer Investigational Site, Montebello, California
  - Pfizer Investigational Site, Monterey Park, California
  - Pfizer Investigational Site, San Francisco, California
  - Pfizer Investigational Site, San Gabriel, California
  - Pfizer Investigational Site, Whittier, California
  - Pfizer Investigational Site, Jacksonville, Florida
  - Pfizer Investigational Site, Jacksonville Beach, Florida
  - Pfizer Investigational Site, Melbourne, Florida
  - Pfizer Investigational Site, Orange Park, Florida
  - Pfizer Investigational Site, Palatka, Florida
  - Pfizer Investigational Site, Saint Augustine, Florida
  - Pfizer Investigational Site, Chicago, Illinois
  - Pfizer Investigational Site, Zion, Illinois
  - Pfizer Investigational Site, Boston, Massachusetts
  - Pfizer Investigational Site, Ann Arbor, Michigan
  - Pfizer Investigational Site, Stony Brook, New York
  - Pfizer Investigational Site, Cleveland, Ohio
  - Pfizer Investigational Site, Corvallis, Oregon
- Canada (3):
  - Pfizer Investigational Site, Edmonton, Alberta
  - Pfizer Investigational Site, Ottawa, Ontario
  - Pfizer Investigational Site, Montreal, Quebec
- Czechia (2):
  - Pfizer Investigational Site, Nový Jičín
  - Pfizer Investigational Site, Prague
- Germany (5):
  - Pfizer Investigational Site, Berlin
  - Pfizer Investigational Site, Essen
  - Pfizer Investigational Site, Frankfurt
  - Pfizer Investigational Site, Freiburg im Breisgau
  - Pfizer Investigational Site, Hamburg
- India (2):
  - Pfizer Investigational Site, Bangalore, Karnataka
  - Pfizer Investigational Site, Pune, Maharashtra
- Italy (4):
  - Pfizer Investigational Site, Napoli
  - Pfizer Investigational Site, Roma
  - Pfizer Investigational Site, Rozzano (Mi)
  - Pfizer Investigational Site, Taormina, ME
- Spain (6):
  - Pfizer Investigational Site, L'Hospitalet de Llobregat, Barcelona
  - Pfizer Investigational Site, Sabadell, Barcelona
  - Pfizer Investigational Site, Girona, Girona
  - Pfizer Investigational Site, Madrid, Madrid
  - Pfizer Investigational Site, Málaga, Malaga
  - Pfizer Investigational Site, Valencia, Valencia
- United Kingdom (4):
  - Pfizer Investigational Site, Southampton, Hampshire
  - Pfizer Investigational Site, Rickmansworth, Middlesex
  - Pfizer Investigational Site, Nottingham, Nottinghamshire
  - Pfizer Investigational Site, Sheffield, Yorkshire

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants who progressed in Docetaxel + Placebo (Phase 2, Double-blind) after consent were eligible to continue to open-label phase. 16 participants crossed-over to open-label phase.
Groups:
- Axitinib + Docetaxel (Phase-1, Lead-in): Axitinib (AG-013736) 5 milligram (mg) tablet orally twice daily (BID) starting from Day 3 of Cycle 1, in cycles of 3 weeks. Docetaxel 80 milligram/square meter (mg/m^2) 1 hour (hr) intravenous (IV) infusion on Day 1 of each cycle, in cycles of 3 weeks.
- Axitinib + Docetaxel (Phase 2, Double-blind): Axitinib (AG-013736) 5 mg tablet orally BID starting from Day 1 of Cycle 1, in cycles of 3 weeks. Docetaxel 80 mg/m^2 1 hr IV infusion on Day 1 of each cycle, in cycles of 3 weeks. Treatment was continued until disease progression, intolerable toxicity, or for 2 cycles after complete response.
- Docetaxel + Placebo (Phase 2, Double-blind): Placebo matched to axitinib (AG-013736) tablet orally BID starting from Day 1 of Cycle 1, in cycles of 3 weeks. Docetaxel 80 mg/m^2 1 hr IV infusion on Day 1 of each cycle, in cycles of 3 weeks. Treatment was continued until disease progression, intolerable toxicity, or for 2 cycles after complete response. Participants with disease progression after consent were continued to open-label phase.
- Axitinib (Phase 2, Open-label): Axitinib (AG-013736) 5 mg tablet orally BID continuously in cycles of 4 weeks.
Period: Phase 1, Lead-in
Arm/Group | Axitinib + Docetaxel (Phase-1, Lead-in) | Axitinib + Docetaxel (Phase 2, Double-blind) | Docetaxel + Placebo (Phase 2, Double-blind) | Axitinib (Phase 2, Open-label)
Started | 6 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0
Not Completed | 6 | 0 | 0 | 0
Not completed — Lack of Efficacy | 4 | 0 | 0 | 0
Not completed — Adverse Event | 1 | 0 | 0 | 0
Not completed — Clinical progression | 1 | 0 | 0 | 0
Period: Phase 2, Double-blind
Arm/Group | Axitinib + Docetaxel (Phase-1, Lead-in) | Axitinib + Docetaxel (Phase 2, Double-blind) | Docetaxel + Placebo (Phase 2, Double-blind) | Axitinib (Phase 2, Open-label)
Started | 0 | 112 | 56 | 0
Treated | 0 | 111 | 56 | 0
Completed | 0 | 0 | 0 | 0
Not Completed | 0 | 112 | 56 | 0
Not completed — Lack of Efficacy | 0 | 59 | 40 | 0
Not completed — Withdrawal by Subject | 0 | 13 | 4 | 0
Not completed — Adverse Event | 0 | 25 | 6 | 0
Not completed — Un-specified | 0 | 14 | 6 | 0
Not completed — Randomized but not treated | 0 | 1 | 0 | 0
Period: Phase 2, Open-label
Arm/Group | Axitinib + Docetaxel (Phase-1, Lead-in) | Axitinib + Docetaxel (Phase 2, Double-blind) | Docetaxel + Placebo (Phase 2, Double-blind) | Axitinib (Phase 2, Open-label)
Started | 0 | 0 | 0 | 16
Completed | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 16
Not completed — Adverse Event | 0 | 0 | 0 | 2
Not completed — Lack of Efficacy | 0 | 0 | 0 | 11
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1
Not completed — Other | 0 | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Axitinib + Docetaxel (Phase 1, Lead-in): Axitinib (AG-013736) 5 mg tablet orally twice daily BID starting from Day 3 of Cycle 1, in cycles of 3 weeks. Docetaxel 80 mg/m^2 1 hr IV infusion on Day 1 of each cycle, in cycles of 3 weeks.
- Docetaxel + Placebo (Double-blind): Placebo matched to axitinib (AG-013736) tablet orally BID starting from Day 1 of Cycle 1, in cycles of 3 weeks. Docetaxel 80 mg/m^2 1 hr IV infusion on Day 1 of each cycle, in cycles of 3 weeks. Treatment was continued until disease progression, intolerable toxicity, or for 2 cycles after complete response. Participants with disease progression after consent were continued with axitinib (AG-013736) 5 mg tablet orally BID continuously in cycles of 4 weeks.
- Total: Total of all reporting groups
Arm/Group | Axitinib + Docetaxel (Phase 1, Lead-in) | Axitinib + Docetaxel (Phase 2, Double-blind) | Docetaxel + Placebo (Double-blind) | Total
Number analyzed (Participants) | 6 | 112 | 56 | 174
Age Continuous [Mean (Standard Deviation); unit: Years] | 50.80 (9.68) | 54.10 (10.43) | 54.70 (10.12) | 54.2 (10.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 112 | 56 | 174
  Male | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Time to Tumor Progression (TTP)
Description: Time in days from start of study treatment to first documentation of objective tumor progression or death due to cancer, whichever comes first. TTP was calculated as first event date minus the date of first dose of study medication plus 1. Tumor progression was determined from oncologic assessment data (where data meet the criteria for progressive disease [PD]).
Time Frame: Phase 2 double-blind baseline until tumor progression or death or discontinuation from study treatment, assessed every 9 weeks up to 129 weeks
Population: Study population included all randomized participants who had a baseline assessment of disease and the correct histological cancer type.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Axitinib + Docetaxel (Phase 2, Double-blind) | Docetaxel + Placebo (Phase 2, Double-blind)
Number analyzed (Participants) | 112 | 55
days | 247 [208 to 265] | 215 [191 to 247]
Statistical Analysis 1: Comparison: Axitinib + Docetaxel (Phase 2, Double-blind) vs Docetaxel + Placebo (Phase 2, Double-blind); P-value was calculated using one-sided Log rank test, stratified for estrogen receptor (ER) status (ER-positive or ER-negative/unknown), prior adjuvant chemotherapy (yes or no), and Eastern Cooperative Oncology Group (ECOG) performance status (less than or equal to [=<1] or 2). The stratified Cox proportional hazards model was fitted, using the same stratification variables as above; Test type: Superiority or Other; p = 0.156, Log Rank; One-sided log-rank test at alpha = 0.1 significance level was used; Hazard Ratio (HR) = 1.237, 95% CI 2-sided [0.819 to 1.867]

2. Secondary Outcome: Percentage of Participants With Objective Response (OR) for Phase 2 (Double-blind)
Description: Percentage of participants with OR based assessment of confirmed complete response (CR) or confirmed partial response (PR) according to Response Evaluation Criteria in Solid Tumors (RECIST). Confirmed responses are those that persist on repeat imaging study at least 4 weeks after initial documentation of response. CR are defined as the disappearance of all lesions (target and/or non target). PR are those with at least 30 percent (%) decrease in the sum of the longest dimensions of the target lesions taking as a reference the baseline sum longest dimensions.
Time Frame: Phase 2 double- blind baseline until the date of first documented progression or discontinuation from the study treatment due to any cause, assessed every 9 weeks up to 129 weeks
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Axitinib + Docetaxel (Phase 2, Double-blind) | Docetaxel + Placebo (Phase 2, Double-blind)
Number analyzed (Participants) | 112 | 55
percentage of participants | 41.1 [31.9 to 50.8] | 23.6 [13.2 to 37.0]
Statistical Analysis 1: Comparison: Axitinib + Docetaxel (Phase 2, Double-blind) vs Docetaxel + Placebo (Phase 2, Double-blind); Test type: Superiority or Other; p = 0.038, Fisher Exact; Difference in response rates = 17.4, 95% CI 2-sided [3.0 to 31.9]

3. Secondary Outcome: Percentage of Participants With Objective Response (OR) for Phase 2 (Open-label)
Description: Percentage of participants with OR based assessment of confirmed complete response (CR) or confirmed partial response (PR) according to Response Evaluation Criteria in Solid Tumors (RECIST). Confirmed responses are those that persist on repeat imaging study at least 4 weeks after initial documentation of response. CR are defined as the disappearance of all lesions (target and/or non target). PR are those with at least 30% decrease in the sum of the longest dimensions of the target lesions taking as a reference the baseline sum longest dimensions.
Time Frame: Phase 2 open-label baseline until the date of first documented progression or discontinuation from the study due to any cause, assessed every 8 weeks up to 58 weeks
Population: All treated (AT) population included participants from Phase 2 who progressed by RECIST criteria while in the placebo + docetaxel treatment group and had a baseline disease assessment and received at least 1 dose of study medication.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Axitinib (Phase 2, Open-label)
Number analyzed (Participants) | 16
percentage of participants | 6.3 [0.2 to 30.2]

4. Secondary Outcome: Duration of Response (DR) for Phase 2 (Double-blind)
Description: Time in days from the first documentation of objective tumor response to objective tumor progression or death due to any cause. Duration of tumor response was calculated as the date of the first documentation of objective tumor progression or death due to cancer minus the date of the first CR or PR that was subsequently confirmed plus 1. DR was calculated for the subgroup of participants with a confirmed objective tumor response.
Time Frame: Phase 2 double-blind baseline until the date of first documented progression or discontinuation from the study due to any cause, assessed every 9 weeks up to 129 weeks
Population: Subgroup of participants from the study population with a confirmed objective tumor response (CR or PR).
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Axitinib + Docetaxel (Phase 2, Double-blind) | Docetaxel + Placebo (Phase 2, Double-blind)
Number analyzed (Participants) | 46 | 13
days | 211 [190 to 276] | 149 [120 to 238]

5. Secondary Outcome: Duration of Response (DR) for Phase 2 (Open-label)
Description: as for outcome 4
Time Frame: as for outcome 3
Population: Subgroup of participants from the AT population with a confirmed objective tumor response (CR or PR).
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Axitinib (Phase 2, Open-label)
Number analyzed (Participants) | 1
days | 1.0 [NA to NA] — 95% confidence interval was not estimable since there was only 1 responder. Hence variability could not be estimated.

6. Other Pre Specified Outcome: Population Pharmacokinetics of Axitinib (AG-013736) for Phase 2 (Double-blind)
Description: Data for this Outcome Measure are not reported here because the analysis population includes participants who were not enrolled in this study. ClinicalTrials.gov is designed for reporting results from only those participants who were enrolled in the study and described in the Participant Flow and Baseline Characteristics modules.
Time Frame: Day 1 (pre-dose), Day 22 and Day 43 and then every 9 weeks up to 129 weeks
Reporting Status: Not Posted
Measure: Mean (Standard Deviation); unit: nanogram/milliliter (ng/mL)

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Groups:
- Axitinib + Docetaxel (Phase-1 Lead-in): Axitinib (AG-013736) 5 mg tablet orally BID starting from Day 3 of Cycle 1, in cycles of 3 weeks. Docetaxel 80 mg/m^2 1 hr IV infusion on Day 1 of each cycle, in cycles of 3 weeks.
Arm/Group | Axitinib + Docetaxel (Phase-1 Lead-in) | Axitinib + Docetaxel (Phase 2, Double-blind) | Docetaxel + Placebo (Phase 2, Double-blind) | Axitinib (Phase 2, Open-label)
Serious Adverse Events (participants affected / at risk) | 1/6 | 54/111 | 17/56 | 2/16
Other Adverse Events (participants affected / at risk) | 6/6 | 111/111 | 56/56 | 12/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Axitinib + Docetaxel (Phase-1 Lead-in) (N=6) | Axitinib + Docetaxel (Phase 2, Double-blind) (N=111) | Docetaxel + Placebo (Phase 2, Double-blind) (N=56) | Axitinib (Phase 2, Open-label) (N=16)
Agranulocytosis (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 9 | 3 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 10 | 3 | 0
Arrhythmia supraventricular (Cardiac disorders) | 0 | 1 | 0 | 0
Left ventricular dysfunction (Cardiac disorders) | 0 | 1 | 0 | 0
Palpitations (Cardiac disorders) | 0 | 1 | 0 | 0
Pericardial effusion (Cardiac disorders) | 0 | 1 | 0 | 0
Restrictive cardiomyopathy (Cardiac disorders) | 0 | 1 | 0 | 0
Angle closure glaucoma (Eye disorders) | 0 | 1 | 0 | 0
Diplopia (Eye disorders) | 0 | 0 | 1 | 0
Uveitis (Eye disorders) | 0 | 1 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 4 | 1 | 0
Duodenal ulcer (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 4 | 2 | 0
Odynophagia (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 1 | 5 | 0 | 0
Volvulus (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 4 | 2 | 0
Asthenia (General disorders) | 0 | 3 | 0 | 0
Chest pain (General disorders) | 0 | 2 | 0 | 0
Haemorrhagic cyst (General disorders) | 0 | 1 | 0 | 0
Mucosal inflammation (General disorders) | 0 | 3 | 0 | 0
Pyrexia (General disorders) | 0 | 6 | 1 | 0
Thrombosis in device (General disorders) | 0 | 1 | 0 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Cholecystitis acute (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Anal abscess (Infections and infestations) | 0 | 1 | 0 | 0
Breast abscess (Infections and infestations) | 0 | 1 | 0 | 0
Bronchopneumonia (Infections and infestations) | 0 | 1 | 0 | 0
Catheter site infection (Infections and infestations) | 0 | 2 | 0 | 0
Clostridial infection (Infections and infestations) | 0 | 1 | 0 | 0
Enterobacter infection (Infections and infestations) | 0 | 1 | 0 | 0
Groin abscess (Infections and infestations) | 0 | 1 | 0 | 0
Herpes zoster (Infections and infestations) | 0 | 0 | 1 | 0
Infection (Infections and infestations) | 0 | 1 | 1 | 0
Influenza (Infections and infestations) | 0 | 0 | 1 | 0
Lower respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 0
Neutropenic sepsis (Infections and infestations) | 0 | 1 | 1 | 0
Oral candidiasis (Infections and infestations) | 0 | 1 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 2 | 0 | 0
Respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 1 | 0
Gamma-glutamyltransferase increased (Investigations) | 0 | 1 | 0 | 0
Neutrophil count decreased (Investigations) | 0 | 1 | 0 | 0
Weight decreased (Investigations) | 0 | 1 | 0 | 0
White blood cell count decreased (Investigations) | 0 | 0 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 4 | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Metastases to meninges (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Metastases to nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Lethargy (Nervous system disorders) | 0 | 1 | 0 | 0
Nervous system disorder (Nervous system disorders) | 0 | 0 | 1 | 0
Radiculopathy (Nervous system disorders) | 0 | 1 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 2 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Nasal septum perforation (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 0 | 0
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Capillary leak syndrome (Vascular disorders) | 0 | 1 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 2 | 0 | 0
Hypertension (Vascular disorders) | 0 | 1 | 0 | 0
Hypotension (Vascular disorders) | 0 | 1 | 0 | 0
Hypothyroidism (Endocrine disorders) | 0 | 0 | 0 | 1
Convulsion (Nervous system disorders) | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Axitinib + Docetaxel (Phase-1 Lead-in) (N=6) | Axitinib + Docetaxel (Phase 2, Double-blind) (N=111) | Docetaxel + Placebo (Phase 2, Double-blind) (N=56) | Axitinib (Phase 2, Open-label) (N=16)
Anaemia (Blood and lymphatic system disorders) | 2 | 10 | 13 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 9 | 0 | 0
Leukopenia (Blood and lymphatic system disorders) | 0 | 15 | 12 | 0
Neutropenia (Blood and lymphatic system disorders) | 4 | 39 | 20 | 0
Conjunctivitis (Eye disorders) | 0 | 15 | 4 | 0
Lacrimation increased (Eye disorders) | 3 | 33 | 11 | 0
Abdominal pain (Gastrointestinal disorders) | 4 | 26 | 5 | 2
Abdominal pain upper (Gastrointestinal disorders) | 0 | 8 | 6 | 2
Constipation (Gastrointestinal disorders) | 2 | 37 | 12 | 2
Diarrhoea (Gastrointestinal disorders) | 5 | 69 | 24 | 4
Dry mouth (Gastrointestinal disorders) | 0 | 9 | 4 | 1
Dyspepsia (Gastrointestinal disorders) | 3 | 16 | 6 | 0
Dysphagia (Gastrointestinal disorders) | 2 | 6 | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 7 | 0 | 0
Glossodynia (Gastrointestinal disorders) | 3 | 8 | 4 | 3
Haemorrhoids (Gastrointestinal disorders) | 1 | 8 | 0 | 0
Nausea (Gastrointestinal disorders) | 5 | 54 | 19 | 10
Oral pain (Gastrointestinal disorders) | 4 | 11 | 5 | 3
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 8 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 3 | 47 | 6 | 1
Vomiting (Gastrointestinal disorders) | 4 | 42 | 17 | 5
Asthenia (General disorders) | 0 | 39 | 10 | 1
Chest pain (General disorders) | 0 | 6 | 7 | 1
Chills (General disorders) | 1 | 8 | 6 | 1
Fatigue (General disorders) | 4 | 52 | 24 | 7
Mucosal inflammation (General disorders) | 3 | 42 | 12 | 1
Oedema peripheral (General disorders) | 1 | 18 | 13 | 1
Pain (General disorders) | 1 | 7 | 9 | 0
Pyrexia (General disorders) | 1 | 22 | 10 | 0
Nasopharyngitis (Infections and infestations) | 0 | 8 | 6 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 7 | 4 | 0
Urinary tract infection (Infections and infestations) | 3 | 14 | 4 | 0
Weight decreased (Investigations) | 2 | 16 | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 3 | 36 | 13 | 5
Dehydration (Metabolism and nutrition disorders) | 4 | 12 | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 6 | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 6 | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 6 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 21 | 10 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 21 | 11 | 2
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 18 | 11 | 2
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 6 | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2 | 10 | 3 | 2
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 2 | 6 | 3 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 | 9 | 5 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 22 | 7 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 6 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 25 | 10 | 6
Dizziness (Nervous system disorders) | 1 | 22 | 6 | 3
Dysgeusia (Nervous system disorders) | 4 | 25 | 10 | 1
Headache (Nervous system disorders) | 3 | 27 | 13 | 6
Hypoaesthesia (Nervous system disorders) | 1 | 9 | 3 | 0
Neuropathy peripheral (Nervous system disorders) | 4 | 14 | 8 | 0
Paraesthesia (Nervous system disorders) | 0 | 13 | 5 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 2 | 16 | 6 | 1
Anxiety (Psychiatric disorders) | 2 | 9 | 5 | 0
Depression (Psychiatric disorders) | 0 | 7 | 4 | 1
Insomnia (Psychiatric disorders) | 0 | 20 | 7 | 0
Dysuria (Renal and urinary disorders) | 1 | 8 | 3 | 0
Pollakiuria (Renal and urinary disorders) | 0 | 7 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 18 | 14 | 2
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 | 10 | 4 | 4
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 23 | 10 | 5
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 | 30 | 10 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 | 20 | 8 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 7 | 5 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 4 | 56 | 30 | 1
Blister (Skin and subcutaneous tissue disorders) | 2 | 7 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 14 | 7 | 2
Erythema (Skin and subcutaneous tissue disorders) | 0 | 9 | 4 | 0
Nail discolouration (Skin and subcutaneous tissue disorders) | 0 | 6 | 0 | 0
Nail disorder (Skin and subcutaneous tissue disorders) | 5 | 23 | 14 | 0
Onycholysis (Skin and subcutaneous tissue disorders) | 0 | 8 | 0 | 0
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 1 | 11 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 13 | 5 | 0
Rash (Skin and subcutaneous tissue disorders) | 2 | 26 | 7 | 2
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 | 10 | 0 | 0
Hypertension (Vascular disorders) | 4 | 36 | 3 | 8
Bradycardia (Vascular disorders) | 1 | 0 | 0 | 1
Tachycardia (Vascular disorders) | 1 | 0 | 3 | 2
Dacryostenosis acquired (Vascular disorders) | 1 | 0 | 0 | 0
Glaucoma (Vascular disorders) | 1 | 0 | 0 | 0
Keratitis (Vascular disorders) | 1 | 0 | 0 | 0
Ocular hyperaemia (Vascular disorders) | 1 | 0 | 0 | 0
Vision blurred (Vascular disorders) | 1 | 0 | 0 | 1
Abdominal discomfort (Vascular disorders) | 2 | 0 | 0 | 1
Dental caries (Vascular disorders) | 1 | 0 | 0 | 0
Flatulence (Vascular disorders) | 2 | 0 | 3 | 0
Haemorrhoidal haemorrhage (Vascular disorders) | 1 | 0 | 0 | 0
Odynophagia (Vascular disorders) | 1 | 0 | 0 | 0
Toothache (Vascular disorders) | 1 | 0 | 4 | 1
Axillary pain (Vascular disorders) | 1 | 0 | 0 | 0
Irritability (Vascular disorders) | 1 | 0 | 0 | 0
Seasonal allergy (Immune system disorders) | 1 | 0 | 0 | 0
Cellulitis (Immune system disorders) | 1 | 0 | 0 | 0
Infected sebaceous cyst (Immune system disorders) | 1 | 0 | 0 | 0
Oral candidiasis (Immune system disorders) | 2 | 0 | 0 | 0
Rhinitis (Immune system disorders) | 1 | 0 | 0 | 0
Tooth abscess (Immune system disorders) | 1 | 0 | 0 | 0
Tooth infection (Immune system disorders) | 1 | 0 | 0 | 0
Vulvovaginal candidiasis (Immune system disorders) | 1 | 0 | 0 | 0
Vulvovaginal mycotic infection (Immune system disorders) | 1 | 0 | 0 | 0
Skin laceration (Immune system disorders) | 1 | 0 | 0 | 0
Alanine aminotransferase (Immune system disorders) | 1 | 0 | 0 | 0
Aspartate aminotransferase (Immune system disorders) | 1 | 0 | 0 | 0
Haemoglobin (Immune system disorders) | 1 | 0 | 0 | 0
Neutrophil count (Immune system disorders) | 1 | 0 | 0 | 0
Neutrophil count decreased (Immune system disorders) | 2 | 0 | 0 | 0
White blood cell count decreased (Immune system disorders) | 2 | 0 | 3 | 0
Hypoalbuminaemia (Immune system disorders) | 1 | 0 | 0 | 0
Pain in jaw (Immune system disorders) | 1 | 0 | 0 | 0
Dyskinesia (Immune system disorders) | 1 | 0 | 0 | 0
Hyperaesthesia (Immune system disorders) | 1 | 0 | 0 | 0
Migraine (Immune system disorders) | 1 | 0 | 0 | 1
Haematuria (Immune system disorders) | 2 | 0 | 0 | 0
Micturition urgency (Immune system disorders) | 1 | 0 | 0 | 1
Urinary incontinence (Immune system disorders) | 1 | 0 | 0 | 0
Vaginal discharge (Immune system disorders) | 1 | 0 | 0 | 0
Vaginal haemorrhage (Immune system disorders) | 2 | 0 | 0 | 0
Vulvovaginal discomfort (Immune system disorders) | 1 | 0 | 0 | 0
Vulvovaginal pain (Immune system disorders) | 1 | 0 | 0 | 0
Nasal congestion (Immune system disorders) | 1 | 0 | 0 | 0
Nasal discomfort (Immune system disorders) | 1 | 0 | 0 | 0
Productive cough (Immune system disorders) | 1 | 0 | 0 | 1
Rhinitis allergic (Immune system disorders) | 1 | 0 | 0 | 0
Sputum discoloured (Immune system disorders) | 1 | 0 | 0 | 0
Upper-airway cough syndrome (Immune system disorders) | 1 | 0 | 0 | 0
Wheezing (Immune system disorders) | 1 | 0 | 0 | 1
Hirsutism (Immune system disorders) | 1 | 0 | 0 | 0
Onychalgia (Immune system disorders) | 1 | 0 | 0 | 0
Pain of skin (Immune system disorders) | 1 | 0 | 0 | 1
Rash erythematous (Immune system disorders) | 1 | 0 | 0 | 0
Skin reaction (Immune system disorders) | 1 | 0 | 0 | 0
Umbilical erythema (Immune system disorders) | 1 | 0 | 0 | 0
Urticaria (Immune system disorders) | 1 | 0 | 0 | 0
Flushing (Immune system disorders) | 1 | 0 | 0 | 0
Hypotension (Immune system disorders) | 1 | 0 | 5 | 1
Eye pain (Immune system disorders) | 0 | 0 | 3 | 0
Abdominal distension (Immune system disorders) | 0 | 0 | 3 | 0
Catheter site pain (Immune system disorders) | 0 | 0 | 4 | 0
Face oedema (Immune system disorders) | 0 | 0 | 4 | 0
Oedema (Immune system disorders) | 0 | 0 | 5 | 0
Dyspnoea exertional (Immune system disorders) | 0 | 0 | 3 | 0
Pleural effusion (Immune system disorders) | 0 | 0 | 5 | 0
Hot flush (Immune system disorders) | 0 | 0 | 4 | 0
Lymphoedema (Immune system disorders) | 0 | 0 | 6 | 0
Lymphadenopathy (Immune system disorders) | 0 | 0 | 0 | 1
Eyelid oedema (Immune system disorders) | 0 | 0 | 0 | 1
Hyperchlorhydria (Immune system disorders) | 0 | 0 | 0 | 1
Oral discomfort (Immune system disorders) | 0 | 0 | 0 | 1
Retching (Immune system disorders) | 0 | 0 | 0 | 1
Catheter site erythema (Immune system disorders) | 0 | 0 | 0 | 1
Chest discomfort (Immune system disorders) | 0 | 0 | 0 | 1
Influenza like illness (Immune system disorders) | 0 | 0 | 0 | 1
Influenza (Immune system disorders) | 0 | 0 | 0 | 1
Sinusitis (Immune system disorders) | 0 | 0 | 0 | 1
Transaminases increased (Immune system disorders) | 0 | 0 | 0 | 1
Flank pain (Immune system disorders) | 0 | 0 | 0 | 1
Groin pain (Immune system disorders) | 0 | 0 | 0 | 1
Muscle fatigue (Immune system disorders) | 0 | 0 | 0 | 1
Balance disorder (Immune system disorders) | 0 | 0 | 0 | 1
Facial neuralgia (Immune system disorders) | 0 | 0 | 0 | 1
Sinus headache (Immune system disorders) | 0 | 0 | 0 | 1
Proteinuria (Immune system disorders) | 0 | 0 | 0 | 1
Postnasal drip (Immune system disorders) | 0 | 0 | 0 | 1
Eczema (Immune system disorders) | 0 | 0 | 0 | 2
Hyperkeratosis (Immune system disorders) | 0 | 0 | 0 | 1

LIMITATIONS AND CAVEATS:
Analysis of TTP (Phase 2, Double-blind) was performed with both discontinuation due to lack of efficacy (LOE) considered a progression and not considered a progression event. Latter was considered primary analysis and former a sensitivity analysis.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.